CLINICAL TRIAL: NCT03082118
Title: Vesair Continued Access Trial: Use of the Vesair® Bladder Control System in the Treatment of Post-Menopausal Female Subjects With Stress Urinary Incontinence
Brief Title: Vesair Continued Access Trial
Acronym: VESICAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solace Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD1007
Record Dates: First submitted 2017-03-11; First posted 2017-03-17 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: All women enrolled are treated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Vesair Arm (Experimental): Subjects treated with the Vesair Bladder Control System at enrollment.
  Interventions: Device: Vesair Bladder Control System

INTERVENTIONS:
Device: Vesair Bladder Control System — Intravesical balloon
  Other Names: Vesair Balloon

SUMMARY:
Single arm study of the Vesair Balloon in postmenopausal women.

DETAILED DESCRIPTION:
All women enrolled will be treated with the vesair balloon and followed for a maximum of 3 years, with balloon replacement annually.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women with SUI or stress predominant mixed incontinence
* Maximum score on IQOL of 60
* Positive cough test for leakage
* Willing to undergo procedures
* Free from infection
* Have previously tried (and failed) noninvasive treatment for SUI

Exclusion Criteria:

* SUI due to SUI
* Urge-predominant mixed incontinence
* Incontinence of neurogenic etiology
* 2 or more UTIs in past year and 1 in past 3 months
* Surgery for SUI in the past 6 months
* taking medication that can be used to treat SUI
* taking medication that affects urinary symptoms for less than 3 months
* undergoing biofeedback
* Grade 3 or worse cystocele
* last menstrual period within 12 months
* oral progesterone or estrogen in the past 12 months
* BMI > 40
* involuntary detrusor contractions or discomfort during bladder filling
* previous stage III or worse cancer
* previous cancer of the urinary tract
* previous symptoms for early stage cancer in the past 2 years
* anticoagulation therapy other than aspirin
* history of prosthetic heart valve
* neurological or connective tissue condition or disease affecting bladder function
* known allergy to device components

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Improvement on patient-reported outcomes | 3-12 months
  Improvement reported on questionnaires

SECONDARY OUTCOMES:
Reduction in leakage events | 3-12 months
  Reduction in leakage events reported on a voiding diary

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Kaiser Permanente Urology, Los Angeles, California
  - Kaiser Permanente Urogynecology, San Diego, California
  - Georgia Center for Women, Atlanta, Georgia
  - Regional Urology, Shreveport, Louisiana
  - Institute for Female Pelvic Medicine and Reconstructive Surgery, Allentown, Pennsylvania
  - Riddle Hospital, Main Line Health, Media, Pennsylvania
  - West Penn Hospital, Allegheny Health Network, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No